Quantitative variables (gestational age, birth weight, age at frenotomy, heart rate pre and post-procedure, increase in heart rate post-procedure, oxygen saturation pre and post-procedure, decrease in oxygen saturation post-procedure, and duration of crying) are described using the mean, standard deviation and range; experimental vs control groups were compared with a Student's t-test. We assessed the equality of variances by using Levene's test and applied the result of the Student's t-test accordingly. Sex, the presence of crying, and adverse effects between the two groups are presented in percentages and compared using Fisher's exact test. Statistical significance was set for a p <0.05. To perform statistical analyses we used STATA version 16.1 (StataCorp, College Station, TX, USA).